CLINICAL TRIAL: NCT01075217
Title: A Phase IV Multi-Center Study to Compare ISOVUE -250 and VISIPAQUE 270 for Motion Artifact and Pain in Peripheral Digital Subtraction Angiography (DSA)
Brief Title: Isovue in Peripheral Digital Subtraction Angiography (DSA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP 119
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2012-04

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Peripheral arterial occlusive disease (PAOD)
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Iopamidol; iodixanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isovue 250 (iopamidol) (Experimental)
  Interventions: Drug: iopamidol
- Visipaque 270 (iodixanol) (Active Comparator)
  Interventions: Drug: iodixanol

INTERVENTIONS:
Drug: iopamidol — Participants received at least one intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
  Other Names: Other name: Isovue 250
  Arms: Isovue 250 (iopamidol)
Drug: iodixanol — Participants received at least one intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
  Other Names: Other name: Visipaque 270
  Arms: Visipaque 270 (iodixanol)

SUMMARY:
No significant differences is expected in observed motion artifacts, heat or pain reported during peripheral DSA performed for diagnostic and/or endovascular therapeutic purposes.

ELIGIBILITY:
Inclusion Criteria:

* provides written informed consent;
* at least 18 years of age;
* scheduled to undergo peripheral DSA for the diagnosis and/or treatment of PAOD

Exclusion Criteria:

* pregnant or lactating female;
* known allergies to one more more ingredients in wither product;
* history of severe congestive heart failure (Class IV);
* previously enrolled or received an investigational compound within 30 days;
* history of hypersensitivity to iodinated contrast agents;
* renal impairment eGFR <60 mL/min/1.73m2, calculated using the MDRD study equation
* any other medical condition decreasing chances of obtaining reliable data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Krix, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: April 2010 (first patient received study agent); Study completion date: December 2011 (final collection date for primary outcome measure) This study was conducted in 6 clinical sites across the United States and 1 in Canada.
Groups:
- Isovue 250; Visipaque 270: Intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Period: Overall Study
Arm/Group | Isovue 250 | Visipaque 270
Started | 84 (88 patients randomized to receive Isovue; 4 of the patients did not meet entry requirements) | 85 (86 patients randomized to receive Visipaque; 1 of the patients did not meet entry requirements)
Completed | 82 | 84
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients who received study agent comprised the baseline population. Four patients assigned to Isovue 250 and 1 assigned to Visipaque 270 did not receive study agent because they did not meet all entry criteria or withdrew before study agent was adminstered
Groups:
- Total: Total of all reporting groups
Arm/Group | Isovue 250 | Visipaque 270 | Total
Number analyzed (Participants) | 84 | 85 | 169
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.77) | 63.1 (8.65) | 63.6 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 54 | 57 | 111
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68 | 71 | 139
  Black or African American | 15 | 13 | 28
  Asian | 1 | 0 | 1
  Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain/Heat in the Lower Extremities Scored by the Participants on the Visual Analog Scale (VAS) Following Intra-arterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA
Description: The 10-centimeter Pain VAS was completed by the Group 1 patients to assess his/her pain level (not scoring heat separately from pain) in the lower extremity of interest. The scale was 0 to 10 cm, with the left end (0 cm)of the scale indicating no pain and the right end (10 cm) of the scale indicating the worst pain.
  The 10-centimeter Pain VAS (excluding Heat assessment, which was separately assessed) was completed by the Group 2 patients to assess his/her pain level in the lower extremity of interest. The scale was 0 to 10 cm, with the left end (0 cm)of the scale indicating no pain and the right end (10 cm) of the scale indicating the worst pain.
  Group 1 completed the Pain VAS (heat not separate from pain). Group 2 completed the Pain VAS for pain only and, separately, the Heat VAS for heat only.
Time Frame: immediately after administration of agent using a power injector for the administration
Population: Patients who received study agent, had the corresponding endpoint evaluations available and had no deviations from the planned protocol were included in the analysis.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Isovue 250 VAS Score Prior to Injection (Baseline); Isovue 250 VAS Score Immediately After Injection; Visipaque 270 VAS Score Prior to Injection (Baseline); Visipaque 270 VAS Score Immediately After Injection: Intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Arm/Group | Isovue 250 VAS Score Prior to Injection (Baseline) | Isovue 250 VAS Score Immediately After Injection | Visipaque 270 VAS Score Prior to Injection (Baseline) | Visipaque 270 VAS Score Immediately After Injection
Number analyzed (Participants) | 77 | 77 | 82 | 82
centimeters
  Group 1 pain and heat not separate (n=42,42,48,48) | 0.6 (1.64) | 3.1 (3.20) | 0.3 (0.87) | 0.7 (1.52)
  Group 2 pain and heat separate (n=35,35,34,34) | 0.4 (1.5) | 1.2 (2.10) | 0.2 (0.77) | 0.8 (1.76)
Statistical Analysis 1: Comparison: Isovue 250 VAS Score Immediately After Injection vs Visipaque 270 VAS Score Immediately After Injection; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value provided is for the difference in pain assessment between Isovue and Visipaque in Group 1, i.e., pain was not assessed separately from heat; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [1.4 to 3.5], Standard Deviation 2.45
Statistical Analysis 2: Comparison: Isovue 250 VAS Score Immediately After Injection vs Visipaque 270 VAS Score Immediately After Injection; Test type: Superiority or Other; p = 0.3244, t-test, 2 sided — P-value provided is for the difference in pain assessment between Isovue and Visipaque in Group 2, i.e., pain was assessed separately from heat; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.5 to 1.4], Standard Deviation 1.94

2. Secondary Outcome: Level of Heat in the Lower Extremities Scored by Group 2 as Assessed on the Heat VAS Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA
Description: The 10-centimeter Heat VAS was completed by the Group 2 patients to assess his/her heat level (separately from pain) in the lower extremity of interest. The scale was 0 to 10 cm, with the left end (0 cm)of the scale indicating no heat and the right end (10 cm) of the scale indicating the worst heat.
  The Heat VAS was completed by the patient before completing the Pain VAS to assess pain.
Time Frame: Immediately after administration of agent using a power injector for the administration
Population: Patients who did not deviate from the planned protocol and had the corresponding endpoint evaluations available were included in the analysis. Group 2 patients provided an assessment of heat by the Heat VAS prior to assessing pain by the Pain VAS.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Visipaque 270 VAS Score Immedicately After Injection: Intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Arm/Group | Isovue 250 VAS Score Immediately After Injection | Visipaque 270 VAS Score Immedicately After Injection
Number analyzed (Participants) | 35 | 34
centimeters | 3.3 (2.57) | 1.7 (2.10)
Statistical Analysis 1: Comparison: Isovue 250 VAS Score Immediately After Injection vs Visipaque 270 VAS Score Immedicately After Injection; Test type: Superiority or Other; p = 0.0059, t-test, 2 sided; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [0.5 to 2.7], Standard Deviation 2.35

3. Secondary Outcome: The Number of Participants With Significant Motion Artifacts (Scores of 3 or 4) Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA.
Description: Using the following 5-point scale, the Investigator reviewed the images for motion artifact in vessels distal to the knee: 0 = None; 1 = Mild, not significant; 2 = Significant, but correctable; 3 = Degrades image quality; 4 = Images uninterpretable. Scores of 3 and 4 were counted as significant motion artifacts.
Time Frame: Immediately postdose
Population: Patients who did not deviate from the planned protocol and had the corresponding endpoint evaluations available were included in the analysis. Patients with significant motion artifact were those with a score of 3 or 4 for motion artifacts in vessels distal to the knee
Measure: Number; unit: participants
Groups:
- Isovue 250 Immediately After Injection; Visipaque 270 Immediately After Injection: Intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Arm/Group | Isovue 250 Immediately After Injection | Visipaque 270 Immediately After Injection
Number analyzed (Participants) | 77 | 82
participants | 2 | 2

4. Secondary Outcome: The Number of Participants Requiring Repeat Injection(s) Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA.
Description: The Investigator assessed the images and recorded the number of repeat power injections required due to motion artifacts for each participant.
Time Frame: Immediately postdose
Population: Patients who did not deviate from the planned protocol and had the corresponding endpoint evaluations available were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Isovue 250 Immediately After Injection | Visipaque 270 Immediately After Injection
Number analyzed (Participants) | 77 | 82
participants | 3 | 1

5. Secondary Outcome: The Number of Participants With Adequate Quality of Opacification Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA
Description: The Investigator assessed all study images obtained for each patient using a 2-point scale (1 = adequate quality; 2 = inadequate quality); assessment was independent of factors or problems relating to the underlying patient condition or the imaging parameters selected.
  Results are provided for patients with adequate quality.
Time Frame: Immediately postdose
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Isovue 250 Quality of Opacification After Injection; Visipaque 270 Quality of Opacification After Injection: Intraarterial injection in one of the following 3 locations: aortic bifurcation (total volume 15-20 mL), iliac arteries (total volume 10-12 mL), or superficial femoral artery (total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Arm/Group | Isovue 250 Quality of Opacification After Injection | Visipaque 270 Quality of Opacification After Injection
Number analyzed (Participants) | 77 | 82
participants | 75 | 82

ADVERSE EVENTS:
Time Frame: Start of investigational product administration through the follow-up period of 1 hour post-injection
Arm/Group | Isovue 250 | Visipaque 270
Serious Adverse Events (participants affected / at risk) | 1/84 | 1/85
Other Adverse Events (participants affected / at risk) | 6/84 | 1/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isovue 250 (N=84) | Visipaque 270 (N=85)
Aortic rupture (Vascular disorders) | 1 (1) | 0 (0) — Procedural event unrelated to study agent
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) — Procedural event unrelated to study agent
Peripheral arterial dissection (Vascular disorders) | 1 (1) | 0 (0) — Procedural event unrelated to study agent
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isovue 250 (N=84) | Visipaque 270 (N=85)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) — Adverse events were reported after the administration of study agent. For 5 patients in the Isovue group and 1 in the Visipaque group, the event of back pain was determined to be procedural, i.e. related to the procedure (e.g., catheter insertion).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. For one site, there is a Clinical Trial Cooperative Research and Development Agreement (CRADA) with a restriction of 180 days after pooled data set is published by the sponsor or 180 after data lock of the complete data.